CLINICAL TRIAL: NCT05557032
Title: Evaluation of the Effectiveness of the Carotid Arteries in Pulse Control Using USG and Manual Palpation Methods in Cardiopulmonary Resuscitation
Brief Title: Pulse Control Using USG and Manual Palpation Methods in Cardiopulmonary Resuscitation
Status: Completed | Type: Observational
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Adnan Yamanoğlu, Assistant professor, Izmir Katip Celebi University
Other Study IDs: 2021-GOKAE-0536
Record Dates: First submitted 2022-09-17; First posted 2022-09-27 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Cardiopulmonary Resuscitation
Keywords: carotid artery; pulse check; Cardiopulmonary Arrest
MeSH Terms: conditions — Heart Arrest | interventions — Cardiopulmonary Resuscitation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: cardiopulmonary resuscitation — pulse checks during cardiopulmonary resuscitation

SUMMARY:
The final approach adopted in Advanced Cardiac Life Support (ACLS) guidelines as defined by the American Heart Association (AHA) and the European Resuscitation Council (ERC) is to minimize the time between chest compressions in cardiopulmonary resuscitation (CPR). Pulse and rhythm checks are recommended between chest compressions and it is stated that this period should not exceed 10 seconds.

All guidelines also state that in cases of low cardiac output or low blood pressure, even if electrocardiographic (ECG) rhythms can be obtained, pulse checks may still fail and an arterial pulse may not be felt during chest compressions. This difficulty in sensing the arterial pulse causes delays in the decision of cardiac arrest in the patient. For this reason, there are cases of cardiac arrest in which the initiation of CPR is delayed or not started at all.

The most common method for checking the pulse is manual palpation. However, since it is an operator-dependent method, it is affected by the experience of the healthcare personnel, the vital values of the patient, and anatomical differences. Therefore, more objective criteria are required to detect a pulse. A clinical study of the reliability of pulse checks showed that most healthcare professionals are unable to detect the presence or absence of a pulse. Another study showed that pulse alone is not sufficient to initiate CPR, and 50% of decisions to initiate CPR based on heart rate are incorrect. Therefore, more objective criteria have been sought to detect the presence of a pulse. For this purpose, evaluations were made regarding the presence of end-tidal carbon dioxide, cardiac echo, and organized rhythm.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (over 18 years of age) with in-hospital or out-of-hospital cardiac arrest

Exclusion Criteria:

* Patients with traumatic arrest
* Conditions affecting carotid pulse palpation and/or USG application (patients with a history of carotid stenosis or dissection, patients undergoing neck surgery, patients with neck abscess hematoma)
* Pregnant arrest patients

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients over 18 years old
Sampling Method: Probability Sample
Enrollment: 536 (Actual)
Dates: Start 2021-12-25 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-09-16 (Actual)

PRIMARY OUTCOMES:
Carotid artery pulse control result using manual and USG in cardiopulmonary resuscitation | 2 minute
  Our aim is to compare the USG and manual methods in evaluating the presence of a pulse during CPR and to determine which method gives the most appropriate time and accuracy.

CONTACTS AND LOCATIONS:
Locations (1):
- IKCU, Atatürk Eğitim ve Araştırma Hastanesi, Acil Tıp, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All data and statistical analyzes will be shared with academics and official institutions requesting the patient's names, provided that they remain confidential, after the permission of the institution.
Supporting Information: Study Protocol, SAP, CSR